CLINICAL TRIAL: NCT05971173
Title: Nutritional Optimization and Bone Health Management for Older Adults Undergoing Hip Fracture Surgery: A Pilot Study
Brief Title: Nutritional Optimization and Bone Health Management for Older Adults Undergoing Hip Fracture Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20230182H
Record Dates: First submitted 2023-07-14; First posted 2023-08-02 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Hip Fractures
Keywords: Older adults; Hip surgery
MeSH Terms: conditions — Hip Fractures | interventions — Geritol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nutritional Supplements (Experimental): Juven and Centrum Silver 50+ will be administered to this group
  Interventions: Drug: Juven; Drug: Centrum Silver 50+
- Control (No Intervention): Standard of care procedures

INTERVENTIONS:
Drug: Juven — Nutritional supplements
  Other Names: Conditionally essential amino acids
  Arms: Nutritional Supplements
Drug: Centrum Silver 50+ — Over the counter nutritional supplement
  Other Names: Multivitamin/multimineral
  Arms: Nutritional Supplements

SUMMARY:
The overall objective of this pilot study is to test a comprehensive nutritional intervention in elderly patients diagnosed with hip fracture, which the study team believe will reduce functional decline, morbidity and mortality.

DETAILED DESCRIPTION:
This collaborative pilot study is led by a PI who is a board-certified orthopaedic surgeon with extensive experience in the care of older adults with hip fractures. In addition, the multidisciplinary study team includes a research health scientist with vast experience in nutrition, preventive health, and gerontology. The study team will also be supported by a physical therapist and researcher in the field of rehabilitation of older adults with musculoskeletal disorders. Furthermore, an occupational therapist with expertise in rehabilitation science, conduct of pilot studies, and analysis of interview data will play an important role in this study. Moreover, the statistical analyses will be performed by an expert statistical consultant from our institution, who will be reimbursed on a fee for service basis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Male or female, aged 65-89 years
3. Closed fracture of the proximal femur including the anatomic areas of femoral neck, intertrochanteric and subtrochanteric region
4. Patient indicated for surgical treatment (surgical fixation or arthroplasty) as per orthopaedic surgeon
5. Ability to take oral medication and be willing to adhere to the study drug regimen and to the nutritional guidance provided by nutritional experts.

Exclusion Criteria:

1. Patients with open fractures
2. Surgical treatment other than surgical fixation or arthroplasty, such as proximal femur resection
3. Known allergic reactions to components of the study drugs or who do not tolerate oral nutritional supplementation (e.g. total parenteral nutrition or food allergies)
4. Decisional impairment
5. Prisoners

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Assessment of surgical complications at 26 weeks | 26 weeks (post surgery)
  Number of subjects that experienced any complications post surgery

SECONDARY OUTCOMES:
Hospital Readmissions | 26 weeks (post surgery)
  Number of hospital re-admissions
Secondary fractures | 26 weeks (post surgery)
  Number of secondary fractures that occurred post surgery
Grip strength | Baseline to 26 weeks
  Change in grip strength from pre- to post-surgery using a hand dynamometer and measured in pounds
Quality of Life Survey (Short-form 36 Health (SF-36)) | Baseline to 26 weeks
  Change in Health related quality of life (QOL) survey, a 36 item survey. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Zelle, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (2):
- United States (2):
  - University Health System, San Antonio, Texas
  - UT Health San Antonio Department of Orthopedics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
All collected deidentified IPD, that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: At the time of publication in a peer reviewed journal